CLINICAL TRIAL: NCT05092620
Title: Adjunct Collection of Additional Biorepository Data From Patients Enrolled in DFC Trials
Brief Title: Adjunct Collection of Additional Biorepository Data From Patients Enrolled in Diabetic Foot Consortium (DFC) Trials
Status: Terminated | Type: Observational
Why Stopped: The Diabetic Foot Consortium studies that fed into the biorepository study were completed (TEWL) and halted prematurely (CMYC), while another DFC study was opened that collected the biospecimens that were previously collected in this study.
Sponsor: University of Michigan (Other)
Collaborators: Indiana University (Other); University of Miami (Other); University of California, San Francisco (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Stanford University (Other)
Responsible Party: Principal Investigator, Cathie Spino, ScD, Research Professor of Biostatistics, SABER Director, University of Michigan
Other Study IDs: HUM00193015; 5U24DK122927-03 (NIH)
Record Dates: First submitted 2021-10-22; First posted 2021-10-25 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes, diabetic foot ulcer, DFU, wound, wound healing
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, urine, wound tissue, wound dressing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Biorepository will guide the Diabetic Foot Consortium (DFC) activities for collection and storing biosamples and data from participants enrolled in other current and future DFC research studies.

DETAILED DESCRIPTION:
Participants enrolling in a parent DFC research study will be concurrently approached about participating in the DFC Biorepository as well. If agreeable, participants will be asked to provide blood, urine, wound debridement tissue and wound dressing samples at the time of enrollment and once more if appropriate and as coincides with the primary study visit schedule. Participants will also be contacted via phone for every six months for two years thereafter to gather longitudinal data about their wound. Data and samples from the Biorepository, along with data collected during the primary study will be available to ancillary researchers.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age > 18 years
* Previous diagnosis of Type 1 or Type 2 diabetes or pre-diabetes per American Diabetes Association (ADA) guidelines
* Inclusion in a part of any planned or approved DFC protocol

Exclusion Criteria:

* An individual who meets exclusion criteria of the primary DFC protocol in which they are enrolled will also be excluded from participation in the biorepository program as well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult diabetic patients with diabetic foot ulcer
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Participants consenting | Up to 2 years
  Proportion of participants consenting to participation in the biorepository from among DFC studies, by study and overall
Biospecimens collected | Up to 2 years
  Proportion of biospecimens collected, by type, from among those expected, by study and overall

CONTACTS AND LOCATIONS:
Overall Officials: Brian Schmidt, DPM, Principal Investigator — University of Michigan; Cathie Spino, ScD, Study Chair — University of Michigan
Locations (5):
- United States (5):
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan